CLINICAL TRIAL: NCT02809508
Title: The Effect of Oily Fish and Poultry on Children's Cardiometabolic Health and Cognitive Function
Acronym: FiSK Junior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Aalborg University Hospital (Other); University of Waterloo (Other)
Responsible Party: Principal Investigator, Camilla Trab Damsgaard, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D218; H-16018225 (Other: The Danish National Committee on Health Research Ethics)
Record Dates: First submitted 2016-06-06; First posted 2016-06-22 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cardiometabolic Health; Cognitive Function
Keywords: Omega-3; Child nutrition; Dietary recommendations; Cardiovascular risk markers; Cognitive function; Mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Poultry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oily fish (Experimental)
  Interventions: Dietary Supplement: Oily fish
- Poultry (control) (Experimental)
  Interventions: Dietary Supplement: Poultry

INTERVENTIONS:
Dietary Supplement: Oily fish — A selection of oily fish, including salmon, herring and mackerel, provided for dinner and lunch
  Arms: Oily fish
Dietary Supplement: Poultry — A selection of poultry, mainly chicken, provided for dinner and lunch
  Arms: Poultry (control)

SUMMARY:
The purpose of FiSK Junior is to investigate whether intake of oily fish compared to poultry affects cardiovascular risk markers, cognitive function, and behaviour in healthy children.

DETAILED DESCRIPTION:
The FiSK Junior study compares the effects of consuming oily fish versus poultry (control) in healthy 8-9 year-old Danish children. The children will be randomized to consume approximately 300 g/week of either oily fish or poultry for 12 weeks. Measurements and biological sampling will be performed at baseline and at the end of the intervention.

The main objective of the study is to investigate the effect on cardiovascular risk markers, primarily blood pressure and plasma triacylglycerol. Moreover, the effects on cognitive function, behaviour, emotions and physiological stress response will be assessed. In addition, change in n-3 long chain polyunsaturated fatty acid status (compliance), anthropometry, body composition, vitamin D status, inflammatory markers, growth markers, physical activity and diet will be measured. Outcomes will be analysed with focus on potential gender- and genotype-specific effects.

ELIGIBILITY:
Inclusion Criteria:

Children must:

* Be 8 - 9 years of age at the start of the intervention
* Be healthy
* Like oily fish and chicken
* Be willing to be randomized to eat fish or chicken
* Not consume oily fish more than once per week 3 months prior to intervention start
* Not consume fish oil 3 months prior to intervention start
* Speak Danish in order to understand the study procedures

Moreover:

* Parents must read and speak Danish, in order to be properly informed about the study procedures
* The child must live in a household with ≤5 persons

Exclusion Criteria:

* Serious chronic illnesses and diseases that may interfere with study outcomes
* Diagnosed Attention Deficit Hyperactivity Disorder (ADHD) or other psychiatric illness
* Intake of medication that may affect study outcomes
* Concomitant participation in other studies involving dietary supplements or blood sampling
* Living in a household with another participating child

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Blood pressure | At 12 weeks
Serum triacylglycerol concentration | At 12 weeks
  Fasting blood level

SECONDARY OUTCOMES:
Serum LDL cholesterol | At 12 weeks
Serum HDL cholesterol | At 12 weeks
Serum insulin | At 12 weeks
Plasma glucose | At 12 weeks
Blood glycosylated haemoglobin (HbA1c) | At 12 weeks
Heart rate | At 12 weeks
BMI z-score | At 12 weeks
Waist circumference | At 12 weeks
Fat mass index by bioimpedance | At 12 weeks
Cognitive function measured by the Cambridge Neuropsychological Test Automated Battery | At 12 weeks
Response inhibition measured by Flanker test | At 12 weeks
Selective attention capacity measured by Stroop Test | At 12 weeks
Attention measured by the D2 Test of Attention | At 12 weeks
Saliva cortisol after cold-pressor task | At 12 weeks
Hair cortisol | At 12 weeks
Compliance measured by content of n-3 long-chain polyunsaturated fatty acids in red blood cells | At 12 weeks

OTHER OUTCOMES:
Behaviour measured by the Strengths and Difficulties Questionnaire | At 12 weeks
  Administered to parent
Behaviour measured by the Behavior Rating Inventory of Executive Function Questionnaire | At 12 weeks
  Administered to parent
Serum insulin-like growth factor-1 | At 12 weeks
Serum C-reactive protein | At 12 weeks
Serum 25-hydroxy-vitamin D | At 12 weeks
Physical activity | At 12 weeks
  Measured by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Camilla T Damsgaard, Assoc Prof, Principal Investigator — University of Copenhagen; Christian Mølgaard, Prof, Study Chair — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Vuholm S, Teisen MN, Molgaard C, Lauritzen L, Damsgaard CT. Sleep and physical activity in healthy 8-9-year-old children are affected by oily fish consumption in the FiSK Junior randomized trial. Eur J Nutr. 2021 Sep;60(6):3095-3106. doi: 10.1007/s00394-021-02490-7. Epub 2021 Jan 30. PMID 33515093
- [Derived] Teisen MN, Vuholm S, Niclasen J, Aristizabal-Henao JJ, Stark KD, Geertsen SS, Damsgaard CT, Lauritzen L. Effects of oily fish intake on cognitive and socioemotional function in healthy 8-9-year-old children: the FiSK Junior randomized trial. Am J Clin Nutr. 2020 Jul 1;112(1):74-83. doi: 10.1093/ajcn/nqaa050. PMID 32529206
- [Derived] Vuholm S, Rantanen JM, Teisen MN, Stark KD, Molgaard C, Christensen JH, Lauritzen L, Damsgaard CT. Effects of oily fish intake on cardiometabolic markers in healthy 8- to 9-y-old children: the FiSK Junior randomized trial. Am J Clin Nutr. 2019 Dec 1;110(6):1296-1305. doi: 10.1093/ajcn/nqz233. PMID 31595295
- [Derived] Damsgaard CT, Lauritzen L, Hauger H, Vuholm S, Teisen MN, Ritz C, Hansen M, Niclasen J, Molgaard C. Effects of oily fish intake on cardiovascular risk markers, cognitive function, and behavior in school-aged children: study protocol for a randomized controlled trial. Trials. 2016 Oct 21;17(1):510. doi: 10.1186/s13063-016-1647-z. PMID 27769289